CLINICAL TRIAL: NCT00534274
Title: Study of Positron Emission Tomography With 3'-Deoxy-3'-[18F] Fluoro-thymidine ([18F]-FLT) for the Evaluation of Response to Neoadjuvant Chemotherapy for Cancers of the Breast
Brief Title: Positron Emission Tomography Using 3'-Deoxy-3'-(18F) Fluorothymidine in Treating Women With Locally Advanced Cancer in One Breast Who Are Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLT01 - UC-0140/0505; FRE-FNCLCC-FLT-01/0505; EU-20754; 2005-005166-37 (EudraCT Number)
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEP FLT (Experimental)
  Interventions: Other: 3'-deoxy-3'-[18F]fluorothymidine

INTERVENTIONS:
Other: 3'-deoxy-3'-[18F]fluorothymidine

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET) using 3'-deoxy-3'-(18F) fluorothymidine, may be effective in assessing the response to chemotherapy before surgery in treating locally advanced breast cancer.

PURPOSE: This clinical trial is studying how well positron emission tomography using 3'-deoxy-3'-(18F) fluorothymidine works in treating women with locally advanced cancer in one breast who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of positron emission tomography (PET) utilizing 3'-deoxy-3'-(18F) fluorothymidine (^18F-FLT) to correctly identify response to neoadjuvant chemotherapy in women with locally advanced unilateral breast cancer.
* Correlate PET-^18F-FLT results with histological response.

Secondary

* Evaluate the correlation of early changes in tumor uptake of ^18F-FLT after the first course of chemotherapy with complete response after treatment completion.
* Evaluate the correlation of early changes in tumor uptake of ^18F-FLT with histologic response in biopsies obtained after 1 course of chemotherapy.
* Determine if the initial intensity of tumor uptake is a predictive value of response to chemotherapy.
* Determine if initial intensity of tumor uptake of ^18F-FLT varies according to histologic type of tumor, indices of proliferation, and tumor cellularity before therapy.
* Determine if the tumor uptake of ^18F-FLT during therapy varies according to histologic type of tumor, indices of proliferation, and tumor cellularity before therapy.
* Evaluate the role of TK1 on the kinetics of ^18 F-FLT.
* Analyze serum.
* Research biomarkers of genomics, transcription, and proteomics.
* Evaluate the toxicity of ^18F-FLT.

OUTLINE: This is a multicenter study.

Patients receive 3'-deoxy-3'-(18F) fluorothymidine (^18F-FLT) IV and undergo positron emission tomography (PET) before the first and second courses of neoadjuvant chemotherapy. Patients receiving bisequential chemotherapy undergo ^18F-FLT-PET before the change in drugs (usually the fourth or fifth course). All patients undergo a final ^18F-FLT-PET after the last chemotherapy course but before surgery.

After completion of study therapy, patients are followed for 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed unilateral breast cancer

  * T2 or T3, any N, M0
  * Unifocal by mammography and ultrasound
* Negative for c-erbB2 by immunohistochemistry (IHC)
* Planning neoadjuvant chemotherapy comprising anthracyclines and/or taxanes, alone or combined
* Measurable disease by ultrasound
* Hormone receptor status not specified

Exclusion criteria:

* Bilateral disease
* Multifocal tumor
* Invasive grade I lobular cancer
* Metastatic disease
* Stage ≥ T4 disease
* Cutaneous invasion, major adherence, or inflammatory disease
* Tumor overexpressing c-erbB2 by IHC (HER 2+++)
* Suspected clinical or radiological lesion (examined or not)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Female
* Menopausal status not specified
* Hematologic, hepatic, and renal function normal
* Not pregnant or nursing
* Fertile patients must use effective contraception

Exclusion criteria:

* Alcohol dependency or prior reaction to ethanol injection
* Impossible to receive study therapy due to geographical, social, or psychological reasons
* Prisoners or patients under supervision

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Participation in another concurrent therapeutic study with an experimental drug

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-11; Primary Completion 2012-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Intensity of tumor uptake of 3'-deoxy-3'-(18F) fluorothymidine (18F-FLT) determined visually and correlated with histological or surgical response according to Sataloff criteria | Post surgery

SECONDARY OUTCOMES:
Intensity of tumor uptake of 18F-FLT by standardized uptake value (SUV) | Post surgery
Variation of tumoral uptake as seen by positron emission tomography (PET) before, during, and after therapy as determined visually and by SUV | Post surgery
Intensity of the tumoral uptake of 18F-FLT on initial exam visually and by SUV | post surgery
Histologic parameters: type, grade, mitotic index, CCIS , and microbiopsy embols after first course of chemotherapy (and on microbiopsy before therapeutic change of sequence in patients receiving bisequential chemotherapy) | post surgery
Immunohistochemical evaluation (estrogen and progesterone receptors, c-erbB2, Ki-67, e-cadherin) | Post-surgery
Rate of thymidine kinase 1 (TK1) | Post surgery
Toxicity by CTC-AE v. 3.0 | Post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Couturier, MD, Study Chair — Centre Hospitalier Regional et Universitaire d'Angers
Locations (24):
- France (24):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Paul Papin, Angers
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hopital Saint Andre, Bordeaux
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Hopital A. Morvan, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Hopital de l'Archet CHU de Nice, Nice
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - CHU Poitiers, Poitiers
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours